CLINICAL TRIAL: NCT04789408
Title: A Phase 1 Open-label, Multicenter Study Evaluating the Safety of KITE-222, an Autologous Anti-CLL-1 CAR T-cell Therapy, in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Study of KITE-222 in Participants With Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to futility
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-486-0201; 2020-000962-40 (EudraCT Number); 2023-507748-35 (Other: European Medicines Agency)
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: KITE-222 (Low Dose) (Experimental): Participants with relapsed or refractory (r/r) acute myeloid leukemia (AML) will receive lymphodepleting chemotherapy (fludarabine and cyclophosphamide) followed by a single infusion of KITE-222 chimeric antigen receptor (CAR) transduced autologous T cells administered intravenously (IV) at a low dose on Day 0 based on participants body weight.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: KITE-222
- Cohort 2: KITE-222 (Higher Dose) (Experimental): Participants with r/r AML will receive lymphodepleting chemotherapy (fludarabine and cyclophosphamide) followed by a single infusion of KITE-222 CAR transduced autologous T cells administered IV at a higher dose on Day 0 based on participants body weight.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: KITE-222
- Cohort 3: KITE-222 (Highest Dose) (Experimental): Participants with r/r AML will receive lymphodepleting chemotherapy (fludarabine and cyclophosphamide) followed by a single infusion of KITE-222 CAR transduced autologous T cells administered IV at the highest dose on Day 0 based on participants body weight.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: KITE-222
- Dose Expansion (Experimental): Participants will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single dose [at the maximum tolerated dose (MTD) determined] of KITE-222.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: KITE-222

INTERVENTIONS:
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously
Biological: KITE-222 — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells administered intravenously

SUMMARY:
The goal of this clinical study is to learn more about the safety and dosing of the study drug, KITE-222, in participants with relapsed/refractory (r/r) acute myeloid leukemia (AML).

ELIGIBILITY:
Key Inclusion Criteria:

* Relapse/refractory (r/r) de novo or secondary acute myeloid leukemia (AML)
* Morphological disease in the bone marrow and/or peripheral blood within 28 days before enrollment
* Prior exposure to the relevant agent class for individuals with AML characterized by a mutation targeted by an approved therapy
* Institutional criteria for allogeneic (allo) - stem cell transplant (SCT) fitness must be met: individuals must have an identified stem-cell donor readily available for potential allo-SCT after therapy with KITE-222
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic status, defined as:

  * Absolute neutrophil count (ANC) ≥ 1000/µL unless, in the opinion of the investigator, cytopenia is due to underlying leukemia
  * Platelet count ≥ 50,000/µL unless, in the opinion of the investigator, thrombocytopenia is due to underlying leukemia
  * Absolute lymphocyte count (ALC) ≥ 100/µL
* Adequate renal, hepatic, pulmonary and cardiac function defined as:

  * Creatinine clearance (as estimated by the Cockcroft Gault formula) ≥ 60 mL/min
  * Serum alanine aminotransferase/aspartate aminotransferase ≤ 2.5 x upper limit of normal
  * Total bilirubin ≤ 1.5 mg/dL, except in individuals with Gilbert's syndrome
  * Cardiac ejection fraction ≥ 50%, no clinically significant pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings
  * Baseline oxygen saturation > 92% on room air and no clinically significant pleural effusion as determined by chest imaging
* Contraception: males and females of childbearing potential must agree to use an effective method of contraception
* Pregnancy testing: females of childbearing potential must have a negative serum or urine pregnancy test

Key Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* Auto-SCT within the 6 weeks before enrollment
* Donor Lymphocyte Infusions (DLI) within 28 days prior to enrollment
* Any drug used for graft-versus-host-disease (GVHD) within 4 weeks prior to enrollment
* Acute GVHD grade II-IV by Mount Sinai Acute GVHD International Consortium criteria
* Active central nervous system (CNS) disease involvement
* Requirement for urgent therapy due to ongoing or impending oncologic emergency (eg, leukostasis or tumor lysis syndrome (TLS)) or the possible requirement for urgent therapy due to ongoing or impending oncologic emergency (eg, spinal cord compression, bowel obstruction, leukostasis, or TLS) at the time of enrollment or KITE-222 infusion
* History of C-type lectin-like molecule-1 (CLL-1)-directed therapy or genetically modified T-cell therapy
* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (eg, cervix, bladder, or breast) unless disease free for at least 3 years after the last definitive therapy
* History of severe hypersensitivity reaction to aminoglycosides
* History of concomitant genetic syndrome associated with bone marrow failure
* Individuals with a genetic syndrome that increases the risk of allo-SCT, including Down syndrome (trisomy 21)
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, atrial fibrillation, or other clinically significant cardiac disease within 12 months before enrollment
* Individuals with cardiac atrial or ventricular leukemia involvement
* History of symptomatic deep vein thrombosis (DVT) or a pulmonary embolism within 6 months of enrollment. History of upper extremity line related DVT within the 3 months of conditioning chemotherapy.
* Primary immunodeficiency disorders
* History of a human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B or C infection
* History of an autoimmune disease resulting in end-organ injury or requiring systemic immunosuppression or systemic disease modifying agents within the last 2 years
* History or presence of a CNS disorder
* Presence or suspicion of a fungal, bacterial, viral, or other infection that is uncontrolled or requiring antimicrobials for management
* Live vaccine received within the ≤ 4 weeks before enrollment, or anticipation of the need for a live vaccination during the course of the study
* Inability to tolerate prophylactic antifungal and antibacterial therapy
* Presence of any indwelling line or drain
* Ongoing Grade 2 or higher toxicities from previous therapies, excluding hematologic toxicities
* Females of childbearing potential who are pregnant or breastfeeding

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (9):
- United States (7):
  - Stanford Cancer Center, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center/James Cancer Hospital, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- France (2):
  - Institut Paoli-Calmettes, Marseille
  - CHU de Toulouse Institut Universitaire du Cancer Toulouse Oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KT-US-486-0201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in France and the United States.
Pre-assignment Details: 17 participants were screened. Dose expansion cohort was not initiated due to early termination of the study. There were no participants enrolled in the expansion cohort.
Groups:
- Cohort 1: KITE-222 (Low Dose): Participants with relapsed or refractory (r/r) acute myeloid leukemia (AML) received lymphodepleting chemotherapy (fludarabine and cyclophosphamide) followed by a single infusion of KITE-222 chimeric antigen receptor (CAR) transduced autologous T cells administered IV at a low dose on Day 0 based on participants body weight.
- Cohort 2: KITE-222 (Higher Dose): Participants with r/r AML received lymphodepleting chemotherapy (fludarabine and cyclophosphamide) followed by a single infusion of KITE-222 CAR transduced autologous T cells administered IV at a higher dose on Day 0 based on participants body weight.
- Cohort 3: KITE-222 (Highest Dose): Participants with r/r AML received lymphodepleting chemotherapy (fludarabine and cyclophosphamide) followed by a single infusion of KITE-222 CAR transduced autologous T cells administered IV at the highest dose on Day 0 based on participants body weight.
Period: Overall Study
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Started | 5 | 3 | 7
Completed | 0 | 0 | 0
Not Completed | 5 | 3 | 7
Not completed — Death | 4 | 3 | 6
Not completed — Did not meet eligibility criteria | 1 | 0 | 0
Not completed — Participant withdrawal of consent from further follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all participants treated with any dose of KITE-222.
Groups:
- Cohort 1: KITE-222 (Low Dose): Participants with r/r AML received lymphodepleting chemotherapy (fludarabine and cyclophosphamide) followed by a single infusion of KITE-222 CAR transduced autologous T cells administered IV at a low dose on Day 0 based on participants body weight.
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose) | Total~(N=12)
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (13.9) | 54 (11.4) | 56 (13.3) | 56 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5
  Male | 2 | 2 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: For Ethnicity, data was not collected for 1 participant in the Cohort 3: KITE-222 (Highest Dose) group.
  Participants
    number analyzed (Participants) | 3 | 3 | 5 | 11
    Hispanic or Latino | 1 | 0 | 0 | 1
    Not Hispanic or Latino | 2 | 3 | 5 | 10
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 2 | 2 | 4 | 8
  Race: Other or More Than One Race | 1 | 1 | 1 | 3
  Race: Black or African American | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 4 | 10
  France | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: DLTs defined as KITE-222-related events with an onset within the first 28 days after the KITE-222 infusion:Grade(GR) 5 event,GR 4 cytokine release syndrome(CRS) or GR 3 CRS not improving to ≤ GR 2 by 72 hours,≥GR 3 cardiac and/or pulmonary event(Exceptions:related to CRS and improve to ≤GR 2 by 72 hours, managed by noninvasive care & resolves to baseline by Day28),GR 4 immune-effector cell-associated neurotoxicity syndrome(ICANS) or other GR 4 adverse events(AEs)associated to neurologic events,GR 3 ICANS(Exceptions: GR 3 ICANS based only on immune-effector cell-associated encephalopathy(ICE) score and/or depressed level of consciousness that improves to ≤GR 2 by 72 hours),≥GR 3 infusion or immediate hypersensitivity reaction,Ongoing GR 4 neutropenia or thrombocytopenia(not due to leukemia persistence)by Day 42 to who have not had conditioning regimen for allo-stem cell transplant,other KITE-222 related GR 3 non-hematologic AEs lasting >7 days,KITE-222-related GR 4 non-hematologic AEs.
Time Frame: Up to 28 days
Population: DLT-evaluable set consisted of participants treated in each dose-escalation cohort who:
  * Received the target dose and were followed for at least 28 days after infusion of KITE-222; or
  * Received a dose of KITE-222 that was lower than the target for that cohort and experienced a DLT during the 28-day post infusion period
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 5
percentage of participants | 0 | 0 | 20

2. Secondary Outcome: Percentage of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical trial participant. The event does not necessarily have a relationship with the study treatment. The definition of an AE includes a worsening of a pre-existing medical condition. Worsening indicates that the pre-existing medical condition has increased in severity, frequency, and/or duration or has an association with a worse outcome. TEAEs were defined as any AEs with onset on or after the date of KITE-222 infusion.
Time Frame: Up to 3.2 months
Population: The Safety Analysis Set consisted of all participants treated with any dose of KITE-222.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants | 100 | 100 | 100

3. Secondary Outcome: Percentage of Participants Who Experienced Laboratory Toxicity Grade Shifts to Grade 3 or Higher Resulting From Increased Parameter Value
Description: Grading categories are determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 1: mild, Grade 2: moderate, Grade 3: severe or medically significant, Grade 4: life-threatening; Grade 5: Death related to AE.
Time Frame: Up to 3.2 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants
  Chemistry: Bilirubin | 0 | 0 | 17
  Chemistry: Direct Bilirubin | 0 | 33 | 33
  Chemistry: Glucose | 33 | 100 | 17
  Chemistry: Alanine Aminotransferase | 0 | 0 | 17
  Chemistry: Alkaline Phosphatase | 0 | 0 | 0
  Chemistry: Aspartate Aminotransferase | 0 | 33 | 17
  Chemistry: Calcium | 0 | 33 | 33
  Chemistry: Potassium | 0 | 0 | 0
  Chemistry: Creatinine | 0 | 0 | 33
  Chemistry: Magnesium | 0 | 0 | 17
  Chemistry: Sodium | 0 | 0 | 0
  Chemistry: Urate | 0 | 0 | 33
  Hematology: Lymphocytes | 0 | 0 | 17

4. Secondary Outcome: Percentage of Participants Who Experienced Laboratory Toxicity Grade Shifts to Grade 3 or Higher Resulting From Decreased Parameter Value
Description: as for outcome 3
Time Frame: Up to 3.2 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants
  Chemistry: Glucose | 0 | 0 | 0
  Chemistry: Albumin | 0 | 0 | 33
  Chemistry: Phosphate | 0 | 67 | 67
  Chemistry: Calcium | 33 | 0 | 33
  Chemistry: Potassium | 33 | 0 | 50
  Chemistry: Magnesium | 0 | 0 | 0
  Chemistry: Sodium | 0 | 0 | 17
  Hematology: Lymphocytes | 100 | 67 | 83
  Hematology: Hemoglobin | 67 | 33 | 50
  Hematology: Leukocytes | 33 | 67 | 67
  Hematology: Platelets | 33 | 0 | 50
  Hematology: Neutrophils | 0 | 33 | 17

5. Secondary Outcome: Time to Neutrophil Recovery
Description: Time to neutrophil recovery after KITE-222 infusion & before the start of the conditioning therapy for allo-SCT was calculated as the time from the date of KITE-222 infusion to the first day when neutrophils are 0.5 × 10^9/liter (L), and as the time from the date of KITE-222 infusion to the first day when neutrophils are 1.0 × 10^9/L. Per European Leukemia Net (ELN) 2017 classification, determined by study investigators, CR was defined as bone marrow (BM) blasts <5%; absence of circulating blasts and blasts with Auer rods;absence of extramedullary disease;absolute neutrophil count (ANC) ≥1.0 × 10^9/L (1000/microliter (μL));platelet count ≥100 × 10^9/L (100000/μL). CRi was defined as all CR criteria except for residual neutropenia (<1.0 × 10^9/L [1000/μL]) or thrombocytopenia (<100 × 10^9/L [100000/μL]).
Time Frame: Up to 3.2 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
months | NA [NA to NA] — None of the participants met the criteria for CR, or Cri, thus the time to neutrophil /platelet recovery could not be calculated. | NA [NA to NA] — None of the participants met the criteria for CR, or Cri, thus the time to neutrophil /platelet recovery could not be calculated. | NA [NA to NA] — None of the participants met the criteria for CR, or Cri, thus the time to neutrophil /platelet recovery could not be calculated.

6. Secondary Outcome: Time to Platelet Recovery
Description: Time to platelet recovery after KITE-222 infusion and before the start of the conditioning therapy for subsequent allo-SCT was calculated as the time from the date of KITE-222 infusion to the first day when platelets are 50 × 10^9/L, and the time from the date of KITE-222 infusion to the first day platelets are 100 × 10^9/L. Per European Leukemia Net (ELN) 2017 classification, determined by study investigators, CR was defined as bone marrow (BM) blasts <5%; absence of circulating blasts and blasts with Auer rods;absence of extramedullary disease;absolute neutrophil count (ANC) ≥1.0 × 10^9/L (1000/microliter (μL));platelet count ≥100 × 10^9/L (100000/μL). CRi was defined as all CR criteria except for residual neutropenia (<1.0 × 10^9/L [1000/μL]) or thrombocytopenia (<100 × 10^9/L [100000/μL]).
Time Frame: Up to 3.2 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
months | NA [NA to NA] — None of the participants met the criteria for CR, or Cri, thus the time to neutrophil /platelet recovery could not be calculated. | NA [NA to NA] — None of the participants met the criteria for CR, or Cri, thus the time to neutrophil /platelet recovery could not be calculated. | NA [NA to NA] — None of the participants met the criteria for CR, or Cri, thus the time to neutrophil /platelet recovery could not be calculated.

7. Secondary Outcome: Composite Complete Remission (CCR) Rate
Description: CCR rate=Percentage of participants who achieve complete remission (CR) + CR without measurable residual disease (CRMRD-) + CR with incomplete hematologic recovery (CRi) per European Leukemia Net (ELN) 2017 classification, determined by study investigators.CR was defined as bone marrow (BM) blasts <5%; absence of circulating blasts and blasts with Auer rods;absence of extramedullary disease;absolute neutrophil count (ANC) ≥1.0 × 10^9/L (1000/microliter (μL));platelet count ≥100 × 10^9/L (100000/μL). CRMRD- if studied pretreatment was defined as CR with negativity for genetic marker by real-time quantitative polymerase chain reaction (RT-qPCR) or CR with negativity by multi-color flow cytometry (MFC).CRi was defined as all CR criteria except for residual neutropenia (<1.0 × 10^9/L [1000/μL]) or thrombocytopenia (<100 × 10^9/L [100000/μL]).
Time Frame: Up to 3.2 months
Population: The participants in the modified intent-to-treat (mITT) analysis set were planned to be analyzed. mITT analysis set were to include all participants enrolled & treated with at least 50% optimal dose of KITE-222 including all participants treated in both dose escalation & dose expansion cohort. Study was discontinued at end of the dose escalation without starting the expansion cohort. Participants in Safety Analysis set were reported.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants | 0 | 0 | 0

8. Secondary Outcome: Overall Remission Rate (ORR)
Description: ORR=percentage of participants who achieved CR+CRMRD- +CRi +morphologic leukemia-free state (MLFS) +partial remission (PR) per the ELN 2017 classification.CR was defined as BM blasts <5%;absence of circulating blasts and blasts with Auer rods;absence of extramedullary disease;ANC ≥1.0 × 10^9/L (1000/ (μL));platelet count ≥100 × 10^9/L (100000/μL).CRMRD- if studied pretreatment = CR with negativity for genetic marker by RT-qPCR or CR with negativity by MFC.CRi was defined as all CR criteria except for residual neutropenia (<1.0 × 10^9/L [1000/μL]) or thrombocytopenia (<100 × 10^9/L [100000/μL]). MLFS=BM blasts <5%;absence of blasts with Auer rods;absence of extramedullary disease;no hematologic recovery required.PR=hematologic criteria of CR decrease of BM blast percentage to 5% to 25%;and decrease of pretreatment BM blast percentage by at least 50%.
Time Frame: Up to 3.2 months
Population: The participants in mITT analysis set were planned to be analyzed. mITT analysis set were to include all participants enrolled & treated with at least 50% optimal dose of KITE-222 including all participants treated in both dose escalation & expansion cohort. Study was discontinued at end of the dose escalation without starting the expansion cohort. Participants in the Safety Analysis Set were reported.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants | 0 | 0 | 16.67

9. Secondary Outcome: Relapse-free Survival (RFS)
Description: For participants who experience CR, CRMRD-, or CRi, RFS was defined as the time between their first CR/CRMRD-/CRi to relapse or death due to any cause. CR was defined as BM blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) ≥1.0 × 10^9/L (1000/μL); platelet count ≥100 × 10^9/L (100000/μL). CRMRD- if studied pretreatment was defined as CR with negativity for a genetic marker by RT-qPCR or CR with negativity by MFC. CR with incomplete hematologic recovery was defined as all CR criteria except for residual neutropenia (<1.0 × 10^9/L [1000/μL]) or thrombocytopenia (<100 × 10^9/L [100000/μL]).
Time Frame: Up to 3.2 months
Population: The participants in the mITT analysis set were planned to be analyzed. mITT analysis set were to include all participants enrolled and treated with at least 50% of the optimal dose of KITE-222 including all participants treated in both the dose escalation cohort and the expansion cohort. The study was discontinued at the end of the dose escalation without starting the expansion cohort. Since no participants experienced CR, CRMRD-, or CRi, RFS could not be evaluated.
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Allogeneic Stem Cell Transplant (Allo-SCT) Rate
Description: The allo-SCT rate was defined as the number of participants who received allo-SCT after being treated with KITE-222 divided by the total number of subjects included in the safety analysis set.
Time Frame: Up to 3.2 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants | 0 | 0 | 0

11. Secondary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the time from the KITE-222 infusion date to earliest date of disease relapse,progressive disease (PD),refractory disease, or death due to any cause.Relapse: Hematologic : BM blasts ≥ 5%,reappearance of blasts, or development of extramedullary disease;Molecular:If studied before treatment, re-occurrence of MRD assessed by RT-qPCR or MFC, PD:Evidence for increase in BM blast percentage and/or increase of absolute blast counts in blood:> 50% increase in marrow blasts over baseline(minimum 15% point increase required with < 30% blasts at baseline or persistent marrow blast > 70%over 3 months without ≥ 100% improvement in ANC to absolute level (> 0.5 × 10^9/L [500/μL], and/or platelet count to > 50 × 10^9/L [50,000/μL] nontransfused); > 50% increase in peripheral blasts(white blood cells (WBC) x % blasts) to > 25 × 10^9/L (>25,000/μL) (absence of differentiation syndrome);New extramedullary disease.Refractory disease:No CR, CRMRD-, or CRi by Week 6 disease assessment.
Time Frame: Up to 12.3 months
Population: The participants in the mITT analysis set were planned to be analyzed. mITT analysis set were to include all participants enrolled and treated with at least 50% of the optimal dose of KITE-222 including all participants treated in both the dose escalation cohort and the expansion cohort. The study was discontinued at the end of the dose escalation without starting the expansion cohort. Participants in the Safety Analysis Set were reported.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
days | 26 [15 to 28] | 23 [9 to 42] | 21.5 [14 to 48]

12. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from KITE-222 infusion to the date of death from any cause.
Time Frame: Up to 12.3 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
months | 2.6 [1.1 to 7.5] | 4.7 [2.9 to 12.3] | 2.6 [0.9 to 6.3]

13. Secondary Outcome: All-cause Mortality Within 30 Days of KITE-222 Infusion
Description: The mortality was calculated by number of deaths, regardless of cause, within 30 days from the KITE-222 infusion date.
Time Frame: Up to 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 1

14. Secondary Outcome: All-cause Mortality Within 60 Days of KITE-222 Infusion
Description: The mortality was calculated by number of deaths, regardless of cause, within 60 days from the KITE-222 infusion date.
Time Frame: Up to 60 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
Participants | 1 | 0 | 3

15. Secondary Outcome: Pharmacokinetics (PK) Parameter: Peak Level of KITE-222 CAR T Cells in Blood
Description: Peak was defined as the maximum number of CAR T cells in blood measured after infusion.
Time Frame: Baseline (Day 0), post dose on Days 3, 7,10, Weeks 2, 3, 4, and 6
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: cells per microliter (cells/µL)
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
cells per microliter (cells/µL) | 2.18 [0.00 to 9.91] | 0.08 [0.00 to 6.05] | 3.88 [0.90 to 79.17]

16. Secondary Outcome: PK Parameter: Area Under the Curve for the Blood Level of KITE-222 CAR T Cells From Day 0 to Day 28 (AUC0-28)
Description: AUC0-28 was defined as the area under curve in a plot of number of CAR T cells against scheduled visit from Day 0 to Day 28.
Time Frame: Baseline (Day 0), post dose on Days 3, 7, 10, Weeks 2, 3, and 4
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: cells/µL*days
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
cells/µL*days | 25.09 [0.00 to 76.90] | 0.47 [0.00 to 58.26] | 26.66 [8.96 to 340.96]

17. Secondary Outcome: Pharmacodynamics (PD) Parameter: Peak Serum Levels of Interferon-gamma (IFNg), Interleukin (IL)-12 P40, IL-10, and IL-15
Description: Peak was defined as the maximum levels of Interferon-gamma (IFNg), Interleukin (IL)-12 P40, IL-10, and IL-15 in serum from baseline to Week 4.
Time Frame: Baseline (Day 0), post dose on Days 1, 3, 5, 7, 9, 11, 13, Weeks 2, 3, 4
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
picograms per milliliter (pg/mL)
  IFNg | 89.80 [20.20 to 463.00] | 150.10 [25.20 to 557.80] | 1876.00 [177.60 to 1876.00]
  IL-12 P40 | 22.30 [21.90 to 339.70] | 195.80 [21.50 to 312.80] | 27.60 [5.70 to 73.00]
  IL-10 | 9.60 [2.20 to 71.50] | 16.50 [12.20 to 34.30] | 145.45 [12.30 to 466.00]
  IL-15 | 30.30 [28.30 to 46.20] | 51.00 [27.00 to 62.70] | 99.65 [24.70 to 185.30]

18. Secondary Outcome: PD Parameter: Peak Serum Levels of IL-2 R Alpha and Ferritin
Description: Peak was defined as the maximum levels of IL-2 R Alpha and Ferritin in serum from baseline to Week 4.
Time Frame: Baseline (Day 0), post dose on Days 1, 3, 5, 7, 9, 11, 13, Weeks 2, 3, 4
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
nanograms per milliliter (ng/mL)
  IL-2 R Alpha | 5.15 [2.92 to 6.71] | 2.90 [2.04 to 6.61] | 21.32 [7.07 to 52.67]
  Ferritin | 16200 [4716.45 to 31600] | 11200 [4539.18 to 17300] | 27900 [5825.07 to 31600]

19. Secondary Outcome: PD Parameter: AUC0-28 for the Serum Levels IFNg, IL-12 P40, IL-10, and IL-15 in Serum
Description: AUC0-28 was defined as the area under curve in a plot of IFNg, IL-12 P40, IL-10, and IL-15 scheduled visit from Day 0 to Day 28.
Time Frame: Baseline (Day 0), post dose on Days 1, 3, 5, 7, 9, 11, 13, Weeks 2, 3, 4
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: pg/mL*days
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
pg/mL*days
  IFNg | 1051.60 [266.55 to 5288.20] | 451.50 [221.55 to 5163.70] | 7317.53 [1161.45 to 20400]
  IL-12 P40 | 575.20 [295.20 to 8040.25] | 1534.05 [433.35 to 5362.45] | 391.60 [216.85 to 1175.30]
  IL-10 | 148.15 [25.35 to 426.30] | 108.95 [59.70 to 401.40] | 809.58 [115.25 to 3078.85]
  IL-15 | 415.15 [382.25 to 1033.70] | 668.60 [181.90 to 1361.60] | 1021.05 [540.55 to 2322.00]

20. Secondary Outcome: PD Parameter: AUC0-28 for the Serum Levels of IL-2 R Alpha and Ferritin
Description: AUC0-28 was defined as the area under curve in a plot of IL-2 R Alpha and Ferritin scheduled visit from Day 0 to Day 28.
Time Frame: Baseline (Day 0), post dose on Days 1, 3, 5, 7, 9, 11, 13, Weeks 2, 3, 4
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: ng /mL*days
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
ng /mL*days
  IL-2 R Alpha | 114.36 [87.00 to 155.16] | 56.61 [43.65 to 145.54] | 302.03 [149.22 to 677.94]
  Ferritin | 208000 [119000 to 353000] | 119000 [86000 to 247000] | 282000 [82900 to 593000]

21. Secondary Outcome: Percentage of Participants Who Develop Anti-KITE-222 CAR Antibodies
Time Frame: Up to 3.2 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to 12.3 months; Adverse Events: Up to 3.2 months
Description: All-cause mortality: The Full Analysis Set consisted of all enrolled participants; Adverse events: The Safety Analysis Set consisted of all participants treated with any dose of KITE-222
Arm/Group | Cohort 1: KITE-222 (Low Dose) | Cohort 2: KITE-222 (Higher Dose) | Cohort 3: KITE-222 (Highest Dose)
All-Cause Mortality (participants affected / at risk) | 4/5 | 3/3 | 7/7
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 4/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: KITE-222 (Low Dose) (N=3) | Cohort 2: KITE-222 (Higher Dose) (N=3) | Cohort 3: KITE-222 (Highest Dose) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Sinusitis fungal (Infections and infestations) | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: KITE-222 (Low Dose) (N=3) | Cohort 2: KITE-222 (Higher Dose) (N=3) | Cohort 3: KITE-222 (Highest Dose) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 2
Facial pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 5
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Bk virus infection (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Epstein-Barr viraemia (Infections and infestations) | 0 | 0 | 1
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3
Sepsis (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viraemia (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Iron overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT04789408/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT04789408/SAP_001.pdf